CLINICAL TRIAL: NCT02416414
Title: Performance Comparison of QuantiFERON Monitor in Solid Organ Transplant Recipients
Status: Terminated | Type: Observational
Why Stopped: Sponsor decided not to go forward with study for FDA submission.
Sponsor: QIAGEN Gaithersburg, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: CST007_10
Record Dates: First submitted 2015-04-07; First posted 2015-04-15 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-03

CONDITIONS: Cell-mediated Immune Response

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Solid Organ Transplant Recipients: Subjects who have received a Solid Organ Transplant.
  Interventions: Device: QuantiFERON Monitor Assay; Device: Existing methodology
- Healthy Controls: Healthy individuals.
  Interventions: Device: QuantiFERON Monitor Assay; Device: Existing methodology

INTERVENTIONS:
Device: QuantiFERON Monitor Assay — Assay to measure cell-mediated immune function using QuantiFERON Monitor assay.
Device: Existing methodology — Assay to measure cell-mediated immune function using existing methodology.

SUMMARY:
To compare the performance of the QuantiFERON Monitor assay against existing methodology.

ELIGIBILITY:
Solid Organ Transplant Recipient

Inclusion Criteria:

* Provide Informed Consent
* Received a solid organ transplant

Exclusion Criteria:

* Pregnancy or recent lactation (<1yr)
* Treatment of Rejection

Healthy Control

Inclusion Criteria:

* Provide Informed Consent

Exclusion Criteria:

* Currently taking any immunomodulatory medication
* A history of immunosuppressive disease or immunosuppression condition or history of autoimmune diseases
* Current pregnancy or recent lactation (<1yr)
* Currently taking antiviral medication
* Currently being treated for infectious diseases

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects who have either received a solid organ transplant or who are healthy.
Sampling Method: Non-Probability Sample
Enrollment: 166 (Actual)
Dates: Start 2015-07; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Cell-mediated immune response. | 1 day (At time of enrollment)

CONTACTS AND LOCATIONS:
Overall Officials: Camille N Kotton, M.D., Principal Investigator — Transplant and Immunocompromised Host Infectious Diseases
Locations (4):
- United States (4):
  - University of California Los Angeles, Los Angeles, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania